CLINICAL TRIAL: NCT06674694
Title: A Phase I Clinical Study of the Safety, Tolerability, and Pharmacokinetics of a Single Dose of Brexpiprazole Long-acting Injection in Healthy Subjects/Patients With Schizophrenia.
Brief Title: The Purpose of This Study is to Determine the Safety, Tolerability, and Pharmacokinetics of Brexpiprazole Long-acting Injection Following a Single Administration in Healthy Subjects/Patients With Schizophrenia.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KL414-3-Ⅰ-01-CTP
Record Dates: First submitted 2024-10-26; First posted 2024-11-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia Disorders
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 20mg dosing group (Experimental): The starting dose is 20 mg and the obtained research results will determine the adjustment of dosage in subsequent study groups.
  Interventions: Drug: Brexpiprazole long-acting injection
- 40mg dosing group (Experimental): The starting dose is 20 mg and the obtained research results will determine the adjustment of dosage in subsequent study groups.
  Interventions: Drug: Brexpiprazole long-acting injection
- 80mg dosing group (Experimental): The starting dose is 20 mg and the obtained research results will determine the adjustment of dosage in subsequent study groups.
  Interventions: Drug: Brexpiprazole long-acting injection
- 160mg dosing group (Experimental): The starting dose is 20 mg and the obtained research results will determine the adjustment of dosage in subsequent study groups.
  Interventions: Drug: Brexpiprazole long-acting injection
- 240mg dosing group (Experimental): The starting dose is 20 mg and the obtained research results will determine the adjustment of dosage in subsequent study groups.
  Interventions: Drug: Brexpiprazole long-acting injection
- 320mg dosing group (Experimental): The starting dose is 20 mg and the obtained research results will determine the adjustment of dosage in subsequent study groups.
  Interventions: Drug: Brexpiprazole long-acting injection

INTERVENTIONS:
Drug: Brexpiprazole long-acting injection — A single injection was administered.

SUMMARY:
Study to evaluate the safety and tolerability of single ascending doses of brexpiprazole long-acting injection in healthy subjects/patients with schizophrenia.

DETAILED DESCRIPTION:
The 20mg group and 40mg group of the study will evaluate the safety and tolerability, PK of single ascending doses of of brexpiprazole long-acting injection in 24 healthy subjects,other groups of the study will evaluate the safety and tolerability, PK of single ascending doses of of brexpiprazole long-acting injection in 32 patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

1. Male and female subjects aged 18 to 65 years (including) at the time of signing the informed consent (the number of single sex in each group is not less than 1/4);
2. Body mass index (BMI) in the range of 19.0-26.0 (including the critical value), and female weight ≥ 45 kg, male weight ≥ 50 kg;
3. Subjects of childbearing potential (including partners) have no pregnancy plan or sperm donation and egg donation plan since signing the informed consent form to within 1 year after the last dose of the investigational drug, and voluntarily take effective contraceptive measures;
4. Sign informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
5. Subjects can communicate well with the investigator, and understand and comply with the requirements of this study.

Patients with schizophrenia:

1. Male and female subjects aged 18 to 65 years (including) at the time of signing the informed consent (the number of single sex in each group is not less than 1/4);
2. Patients diagnosed with schizophrenia according to ICD-10, and the positive and negative symptom scale (PANSS) score ≤ 70 points, and the investigator judged stable disease within 4 weeks before screening;
3. Body mass index (BMI) ≥ 18.5 kg/m2 and < 35.0 kg/m2, and female weight ≥ 45 kg, male weight ≥ 50 kg;
4. Subjects need to complete the tolerance test according to the protocol requirements;
5. Subjects of childbearing potential (including partners) have no pregnancy plan or sperm donation and egg donation plan since signing the informed consent form to within 1 year after the last dose of the investigational drug, and voluntarily take effective contraceptive measures;
6. Subjects and their guardians signed informed consent;
7. Subjects and their guardians agree to comply with the protocol and cooperate with the investigator to complete the trial.

Exclusion Criteria:

Healthy Volunteers:

1. History of cardiovascular system (such as history of ischemic heart disease), endocrine system, urinary system, nervous system, hematology, immunology (including personal or family history of hereditary immunodeficiency), metabolic abnormalities, and the researchers believe that there is still clinical significance;
2. Physical examination, vital signs, 12-lead electrocardiogram, clinical laboratory tests (including hematology, urinalysis, serum biochemistry, thyroid panel, coagulation panel, serum prolactin, virological examination, lipid panel, serum pregnancy test (only women of childbearing age) and glycosylated hemoglobin, etc.), chest X-ray or CT and B-ultrasound with Injection site results in injection site are abnormal and clinically significant;;
3. Those who have taken any brexpiprazole preparation within 28 days prior to oral tolerance test drugs (brexpiprazole tablets);
4. Those who have been enrolled in clinical trials of brepiprazole long-acting injection and have received the test drug administration;
5. Participate in any drug or medical device clinical trial and receive the treatment of the investigational drug or medical device within 28 days before dosing (other than the drug/equipment used in this study), except for subjects participating in the research or observational study;
6. Those who have used any drugs that interact with brepiprazole within 30 days before administration [including CYP3A4 inducers and inhibitors, CYP2D6 inducers and inhibitors] (except topical preparations with local effects);
7. Those who have used any drugs within 14 days before administration [including prescription drugs, over-the-counter drugs, traditional Chinese medicine, etc.] (except topical preparations with local effects);
8. Consumption of foods or beverages rich in xanthine (such as sardines, animal liver, etc.), grapefruit (such as grapefruit, western grapefruit, lime, carambola, etc.), caffeine (such as coffee, strong tea, cola, milk tea, etc.) within 48 hours before dosing, or other special diet that can affect drug absorption, distribution, metabolism and excretion;
9. Those who drink excessive amounts (more than 8 cups, 1 cup = 250 mL) of tea or coffee or beverages rich in xanthine/caffeine/grapefruit (such as milk tea, cola, fruit juice, etc.) before administration;
10. Previous alcohol abuse (i.e., men drink more than 28 standard units per week, women drink more than 21 standard units per week (1 standard unit contains 14 g alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine), or frequent alcohol consumption within the first 6 months before screening (more than 14 standard units per week) and determined by the investigator to affect the test, or unwilling to stop drinking or any alcohol-containing products from the date of screening to the last PK blood collection period;
11. Those who smoke more than 3 cigarettes per day within 3 months before dosing, or are unwilling to stop using any tobacco products from the date of screening to the last PK blood collection in the trial;
12. Those with a history of drug dependence or a history of drug abuse;
13. Positive urine drug abuse screening;
14. Alcohol breath test positive;
15. Those who donate blood or transfuse blood products or use blood products within 1 month before administration (> 200 mL);
16. Those who have undergone surgery within 1 month before administration, or who plan to undergo surgery from the date of screening to the last PK blood collection period of the trial;
17. Those who are allergic or allergic to any component of this product and excipients (allergic to two or more drugs or food);
18. History of needle sickness or blood sickness with clinical significance judged by the investigator to;
19. Pregnant or lactating women;
20. Those who have unprotected sex within 2 weeks prior to administration;
21. The investigator judged that it was not suitable to participate in this trial.

Patients with schizophrenia:

1. Patients with other psychiatric diseases other than schizophrenia diagnosed according to ICD-10 (except the diagnosis of concomitant symptoms of schizophrenia);
2. Participate in any drug or medical device clinical trial and receive the treatment of the investigational drug or medical device within 28 days before dosing (other than the drug/equipment used in this study), except for subjects participating in the research or observational study;
3. Those who have taken any brexpiprazole tablets for tolerance testing within 28 days prior to oral tolerance test drugs (brexpiprazole tablets);
4. Those who have been enrolled in the clinical trial of brexpiprazole long-acting injection and received the test drug administration;
5. More than 1 other antipsychotic drug was used before administration (except for the brexpiprazole tablets given for tolerance testing, which can be combined with ≤ 1 other antipsychotic drug and the drug has been treated at a stable dose for ≥ 14 days before administration);
6. Those who have received other antipsychotic long-acting injection treatment and the interval from the first dose is shorter than that of the long-acting injection;
7. Patients with clinically significant cardiovascular and cerebrovascular diseases, including but not limited to: Concomitant cardiac insufficiency, Severe arrhythmias requiring treatment, Ischemic heart disease requiring treatment, Previous or current congenital heart disease, Previous or present severe organic heart disease, History of stroke or transient ischemic attack within 1 year prior to screening, QTc interval ≥ 450 ms in men or ≥ 470 ms in women, Orthostatic hypotension (decrease in systolic blood pressure (SBP) ≥ 20 mmHg or diastolic blood pressure (DBP) ≥ 10 mmHg within 3 minutes after changing from supine to upright position), Heart rate < 50 bpm or > 100 bpm at rest, Uncontrolled hypertension (SBP > 160 mmHg and/or DBP > 100 mmHg);
8. Patients with poorly controlled diabetes (HbA1c ≥ 7.0%);
9. Pre-dose hematopoiesis and major organ function indicators meet any of the following criteria: White blood cell count < 3.0 × 109/L, neutrophil count < 1.5 × 109/L, platelet count < 75 × 109/L, red blood cell count < 3.0 × 1012/L, hemoglobin < 100 g/L;Total bilirubin > 2 times the upper limit of normal, alanine aminotransferase > 2 times the upper limit of normal, and aspartate aminotransferase > 2 times the upper limit of normal;Creatinine > 1.5 times the upper limit of normal;Creatine kinase > 3 times the upper limit of normal;
10. Previous alcohol abuse (i.e., men drink more than 28 standard units per week, women drink more than 21 standard units per week (1 standard unit contains 14 g alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine), or frequent alcohol consumption within the first 6 months before screening (more than 14 standard units per week) and determined by the investigator to affect the test, or unwilling to stop drinking or any alcohol-containing products from the date of screening to the last PK blood collection period;
11. Those who drink excessive amounts (more than 8 cups, 1 cup = 250 mL) of tea or coffee or beverages rich in xanthine/caffeine/grapefruit (such as milk tea, cola, fruit juice, etc.) before administration;
12. Those who smoke more than 3 cigarettes per day within 3 months before dosing, or are unwilling to stop using any tobacco products from the date of screening to the last PK blood collection in the trial;
13. Alcohol breath test positive;
14. Those with a history of drug dependence or a history of drug abuse;
15. Positive urine drug abuse screening;
16. Those who donate blood or transfuse blood products or use blood products within 1 month before administration (> 200 mL);
17. Those who have undergone surgery within 1 month before dosing, or who plan to undergo surgery from the date of screening to the last PK blood collection period of the trial;
18. Patients with Parkinson's disease, malignant syndrome or dementia-related psychosis;
19. Previous or current tardive dyskinesia (the 8th item score of the involuntary movement scale (AIMS) ≥ 3) or severe akathisia (BARS) overall clinical assessment score of 5 points;
20. Patients with epilepsy or convulsive diseases (except febrile convulsions);
21. Subjects with severe suicidal tendency: the fourth and fifth items of "suicidal ideation" in the Columbia Suicide Severity Rating Scale (C-SSRS) answered "Yes" and the most recent episode within 6 months met the criteria;Or any one of the "suicidal behavior" in the C-SSRS answered "yes" and the most recent episode within 2 years met any of the 5 items;Or, in the opinion of the investigator, the subject is at serious risk of suicide;
22. Have a history of needle sickness or blood sickness, and judged by the investigator to have clinical significance;
23. Those who are allergic or allergic to any component of this product and excipients (allergic to two or more drugs or food);
24. Those who have received electroconvulsive therapy within 14 days prior to screening;
25. Positive for HBsAg, HCV-Ab, Anti-HIV, syphilis antibody;
26. Pregnant or lactating women;
27. Those who have unprotected sex within 2 weeks prior to dosing;
28. Those who have used the following drugs or food before administration: Received any prescription of traditional Chinese medicine preparations, including traditional Chinese medicine, Chinese herbal decoction pieces, Chinese patent medicine, etc., within 14 days (except topical preparations with local effects), Treatment with CYP3A4 or CYP2D6 inhibitors or inducers within 7 days or 5 drug half-lives, whichever is longer (except topical preparations with local effects), Consumption of foods or beverages rich in xanthine (e.g., sardines, animal liver, etc.), grapefruit (e.g., grapefruit, grapefruit, lime, carambola, etc.), caffeine (e.g. coffee, strong tea, cola, milk tea, etc.), or other special diet that can affect drug absorption, distribution, metabolism and excretion within 48 hours;
29. The investigator judged that it was not suitable to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of reported Adverse Events (AE) | Collected from signing of informed consent until 90 days after a single dose.
  Safety and tolerability was assessed by the number of participants with adverse events (AE).
Clinical Laboratory Tests | Collected from signing of informed consent until 90 days after a single dose.
  Hematology, Serum chemistry, Lipid Panel, Glycated Hemoglobin, Urinalysis, Coagulation Panel will be performed.
Change in physical exam results | Collected from signing of informed consent until 90 days after a single dose.
  Investigator will perform complete physical exam and document any clinically significant conditions. Body height and weight will also be measured for BMI calculation and weight will be measured as part of all subsequent physical exams.
Vital signs | Collected from signing of informed consent until 90 days after a single dose.
  Vital signs include respiration, temperature, pulse, and blood pressure.
ECG Reading | Collected from signing of informed consent until 90 days after a single dose.
  12-lead ECG include heart rate, ventricular rate, RR interval, PR interval, QRS duration and QT intervals will be recorded.
Extrapyramidal Symptoms (EPS) Rating Scale | Collected from signing of informed consent until 90 days after a single dose.
  SAS, AIMS , BARS will be assess by trained trial center staff [Only patients with schizophrenia].
Change in Suicidality via Columbia-Suicide Severity Rating Scale | Collected from signing of informed consent until 90 days after a single dose.
  Baseline version and Since Last Visit version of CSSRS will be completed by trained trial center staff [Only patients with schizophrenia].
Injection site assessment | Collected from signing of informed consent until 90 days after a single dose.
  Injection site will be assessed by Investigator.Which includes pain, swelling, redness, induration, etc.

SECONDARY OUTCOMES:
Maximum peak plasma concentration (Cmax) [Pharmacokinetics] | 90 days after a single dose.
  Samples will also be collected until 90 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .
Time of Cmax (tmax) [Pharmacokinetics] | 90 days after a single dose.
  Samples will also be collected until 90 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .
Area under the concentration-time curve (AUC) from time zero to time "t" [Pharmacokinetics] | 90 days after a single dose.
  Samples will also be collected until 90 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .
AUC from time zero to infinity (AUC∞) [Pharmacokinetics] | 90 days after a single dose.
  Samples will also be collected until 90 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .
Terminal-phase elimination half-life (t1/2,z) [Pharmacokinetics] | 90 days after a single dose.
  Samples will also be collected until 90 days after a single dose(samples will be collected in the morning). PK parameters will be assessed for plasma brexpiprazole and its metabolite(s) .

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anding Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No